CLINICAL TRIAL: NCT01070589
Title: The Effect of Obesity on Growth Hormone Response to Anaerobic Exercise
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC01922009CTIL
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Obesity
Keywords: Obesity; Growth hormone secretion; Anaerobic exercise
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Obese: BMI>30
- Group 2: control: Group 2:Normal weight (BMI <25). age and gender matched.

SUMMARY:
The aim of the present study is to asses the effect of obesity on anaerobic exercise's growth hormone (GH) response.

DETAILED DESCRIPTION:
Exercise is a potent physiological stimulator of growth hormone (GH) release. GH is an important factor in the distribution of fat and lean tissue in the body. Previous studies suggested that the GH response to aerobic exercise may be attenuated by obesity. The effect of obesity on GH response to anaerobic effort is unclear. The aim of the present study is to asses the effect of obesity on anaerobic exercise's GH response. We will recruit 12 obese (BMI > 30) healthy adults and 12 age and gender matched normal weight (BMI < 25) controls. All the participants will conduct a "wingate" anaerobic test (30 seconds of intense effort against resistance calculated by the individual's body weight). Blood sample for GH level will be collected at 5 different time (0, 20, 30, 40 and 60 minutes after the test). We will compare the GH response in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female
* Age 18-40

Exclusion Criteria:

* Male
* Age <18, >40
* Heart, Liver, Kidney or Hypophyseal disease
* Medications that may alter GH secretion (eg Steroids, Eltroxin)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy female Age 18-40 years
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Allon Eliakim, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel